CLINICAL TRIAL: NCT00187863
Title: Biopsychosocial Factors' Influence on Shoulder Pain
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 61-2005
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Exercise induced pain perception
  Interventions: Behavioral: pain perception
- Surgical pain perception
  Interventions: Behavioral: pain perception

INTERVENTIONS:
Behavioral: pain perception — pain perception

SUMMARY:
The purpose of this study is to determine which factors are associated with the development of chronic shoulder pain and disability.

DETAILED DESCRIPTION:
The purpose of this study is to determine which factors are associated with the development of chronic shoulder pain and disability. Previous studies have suggested that specific genes influence pain perception. Other studies have suggested that specific psychological factors influence pain perception. We plan to investigate both of these factors to see if they contribute to the development of chronic shoulder pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* chronic shoulder pain and disability

Exclusion Criteria:

* none

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic shoulder pain and disability
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2005-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Disability | Baseline to 12 months
  Measurement using the quick DASH
Pain intensity | Baseline to 12 months
  Measured by the Brief Pain Inventory

SECONDARY OUTCOMES:
Physical impairment | Baseline to 12 months
  Measured shoulder range of motion
Activity evoked pain | Baseline to 12 months
  Measured by Numerical Rating Scale with shoulder movement

CONTACTS AND LOCATIONS:
Overall Officials: Steven Z. George, PT, Ph.D., Principal Investigator — University of Florida
Locations (1):
- UF Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States

REFERENCES:
- [Derived] George SZ, Wu SS, Wallace MR, Moser MW, Wright TW, Farmer KW, Greenfield WH 3rd, Dai Y, Li H, Fillingim RB. Biopsychosocial Influence on Shoulder Pain: Influence of Genetic and Psychological Combinations on Twelve-Month Postoperative Pain and Disability Outcomes. Arthritis Care Res (Hoboken). 2016 Nov;68(11):1671-1680. doi: 10.1002/acr.22876. Epub 2016 Oct 6. PMID 26945673